CLINICAL TRIAL: NCT01767012
Title: Aqueous Flare of a Hydrophobic Acrylic Single-piece Open-loop IOL With Modified Material Surface Properties
Acronym: POL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, MD, MBA, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Viros_POLYLENS
Record Dates: First submitted 2013-01-06; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Cataract; Diabetes; Pseudoexfoliation Syndrome
MeSH Terms: conditions — Cataract; Diabetes Mellitus; Exfoliation Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Polylens EC-Y10-PAL (uncoated) (Active Comparator): hydrophobic acrylic IOL (no coating) implantation during cataract surgery
  Interventions: Device: Polylens EC-Y10-PAL (uncoated)
- Polylens EC-Y10H-PAL (coated) (Active Comparator): hydrophobic acrylic heparin-coated IOL implantation during cataract surgery
  Interventions: Device: Polylens EC-HY10-PAL (coated)

INTERVENTIONS:
Device: Polylens EC-HY10-PAL (coated) — hydrophobic acrylic IOL with modified surface properties (Heparin-coating)
  Arms: Polylens EC-Y10H-PAL (coated)
Device: Polylens EC-Y10-PAL (uncoated)
  Other Names: hydrophobic acrylic IOL
  Arms: Polylens EC-Y10-PAL (uncoated)

SUMMARY:
Modern phacoemulsification techniques have made cataract surgery safe and efficient over the past several decades. Although the phacoemulsification procedure has improved greatly, cataract surgery still involves trauma. One of the surgical traumas during cataract surgery is the direct trauma of the anterior uvea, resulting in a later chronic immune reaction of the uvea to the implanted intraocular lens (IOL). 1 The breakdown of the blood-aqueous barrier (a measure of the uveal reaction) clinically presents as flare in the anterior chamber. 2 Petternel et al. 3 explained that the protein content of the aqueous humor may mainly arise from the iris root and iris vessels in the anterior chamber. The peak of this flare and cell intensity in the anterior chamber was shown to be reached during the first two days after cataract surgery 4 and flare levels were back to the preoperative values about one year after cataract surgery. 5, 6 Influencing factors are surgical technique 7, perioperative treatment 8, IOL biomaterial and design 9 and host reaction to the IOL.

In this study the otherwise same IOL concerning material and design, but one with a new surface modification will be compared to assess the influence on aqueous flare and cell intensity in the anterior chamber. The Polylens (Polytech, Rossdorf, Germany) is a hydrophobic acrylic single-piece open-loop IOL and is available with the standard surface and a novel modified surface.

To assess the efficacy of the newly modified surface of the Polylens IOL compared to the same IOL without a modified surface concerning flare and cell intensity in the anterior chamber as well as cellular components on the IOL surface and lens epithelial out-growth from the rhexis after cataract surgery in eyes of patients with diabetes mellitus and pseudoexfoliation syndrome, which typically have a higher incidence of post-operative intra-ocular inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract
* Age 40 and older
* Diabetes mellitus OR pseudoexfoliation syndrome

Exclusion Criteria:

* Preceding ocular surgery or trauma

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Amount of aqueous flare measured with a Laser flare meter | 1 hour - 3 months postoperatively
  The amount of aqueous flare was measured with a Laser flare meter (Kowa FM-600, Kowa Optimed, USA).The unit of measurement is photon counts per millisecond (pc/ms). The higher flare values, the higher the intracameral amount of protein and, therefore, the higher the intraocular inflammatory response.

SECONDARY OUTCOMES:
Anterior capsule opacification (measured as brightness of anterior capsular reflect on slitlamp photographs) | 1 hour to 3 months postoperatively
  Objective ACO evaluation was obtained after taking 2 slit lamp images in a standardised way of each eye: the area of the anterior capsule in contact with the IOL was defined as the area of interest. Part of the dark area not directly illuminated by the slit beam within the capsulorhexis served as the control area. The difference in brightness between the area of interest and the control area defined the grade of fibrosis in per cent, with 0% representing a clear anterior capsule and 100%, a completely white anterior capsule.

OTHER OUTCOMES:
IOL centration measured with a Purkinje-meter | 3 months post-OP
  The amount of IOL decentration (mm) was measured with a Purkinje-meter system, which analyses misalignment of the optical surfaces of the eye due to position of Purkinje-reflexes.
IOL tilt measured with a Purkinje-meter | 3 months postOP
  The amount of IOL tilt (°) was measured with a Purkinje-meter system, which analyses misalignment of the optical surfaces of the eye due to position of Purkinje-reflexes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanusch-Krankenhaus, Vienna, Vienna, Austria